CLINICAL TRIAL: NCT07090577
Title: Serial Multiomics Profiling Using Serum and Cerebrospinal Fluid Samples Following Out-of-hospital Cardiac Arrest: a Prospective Observational Study
Brief Title: Multiomics Profiling of CSF in Cardiac Arrest Survivors
Acronym: MOPCAS
Status: Active, not recruiting | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Changshin Kang, Assistant professor, Chungnam National University Hospital
Other Study IDs: CNUH-202507010; RS-2025-00554697 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest (CA); Hypoxic-Ischemic Brain Injury; Post-Resuscitation Syndrome
Keywords: cardiac arrest; hypoxic-ischemic brain injury; post-resuscitation syndrome; multiomics; cerebrospinal fluid
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good neurologic outcome: Cerebral Performance Category (CPC) : 1 or 2
- poor neurologic outcome: Cerebral Performance Category (CPC) : 3 to 5

SUMMARY:
The goal of this observational study is to identify further pathophysiologic mechanism of secondary brain injury following cardiac arrest by using serial multiomics profiling of serum and cerebrospinal fluid (CSF) samples. The main question it aims to answer is:

A. The main question it aims to answer is: What are the dynamic molecular changes in serum and CSF that reflect the pathophysiological mechanisms of secondary brain injury after cardiac arrest? B. What are the differences in serum and CSF multiomic signatures between varying severities of cardiac arrest, and how are these differences associated with the underlying pathophysiological mechanisms of secondary brain injury?

Serum and CSF samples that have already been prospectively collected from participants and stored in the BioBank will be used for this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Out-of-hospital cardiac arrest (OHCA)
* Patients who have received post-resuscitation care including temperature control due to unconsciousness (Glasgow Coma Score < 8) after sustained ROSC.
* Patients who consented to the placement of lumbar catheter for storing cerebrospinal fluid and blood samples in a human biobank.

Exclusion Criteria:

* Patients diagnosed with a central nervous system-related disease before cardiac arrest
* Patients who have undergone extracorporeal circulatory membrane oxygenation therapy
* Patients who died within 24 hours from post-resuscitation care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an out-of-hospital cardiac arrest who underwent post-resuscitation care
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome | after 6 months from return of spontaneous circulation
  Cerebral Performance Category (CPC) score

SECONDARY OUTCOMES:
The Pittsburgh Cardiac Arrest Category (PCAC) | immediately after return of spontaneous circulation
  Illness severity of cardiac arrest

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to ethical and privacy concerns. However, data sharing may be possible upon reasonable request with prior approval from the ethics committee and the principal investigator

REFERENCES:
- [Background] You Y, Park JS, Min JH, Jeong W, Ahn HJ, In YN, Jeon SY, Lee JK, Kang C. Blood-brain barrier permeability for the first 24 hours in hypoxic-ischemic brain injury following cardiac arrest. Resuscitation. 2024 May;198:110150. doi: 10.1016/j.resuscitation.2024.110150. Epub 2024 Feb 23. PMID 38401708
- [Background] Stopa V, Lileikyte G, Bakochi A, Agarwal P, Beske R, Stammet P, Hassager C, Arman F, Nielsen N, Devaux Y. Multiomic biomarkers after cardiac arrest. Intensive Care Med Exp. 2024 Sep 27;12(1):83. doi: 10.1186/s40635-024-00675-y. PMID 39331333
- [Background] Lileikyte G, Bakochi A, Ali A, Moseby-Knappe M, Cronberg T, Friberg H, Lilja G, Levin H, Arman F, Kjellstrom S, Dankiewicz J, Hassager C, Malmstrom J, Nielsen N. Serum proteome profiles in patients treated with targeted temperature management after out-of-hospital cardiac arrest. Intensive Care Med Exp. 2023 Jul 17;11(1):43. doi: 10.1186/s40635-023-00528-0. PMID 37455296